CLINICAL TRIAL: NCT05688423
Title: Integrated Care and Treatment for Severe Infectious Diseases and Substance Use Disorders Among Hospitalized Patients
Acronym: CTN0121
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: University of Miami (Other); Emory University (Other); National Institute on Drug Abuse (NIDA) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Principal Investigator, Lisa Metsch, Dean of Columbia University School of General Studies, Professor in Department of Sociomedical Sciences, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20221134; UG1DA013720 (NIH)
Record Dates: First submitted 2022-11-21; First posted 2023-01-18 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Injection Site Infection; Substance Use Disorders
Keywords: substance use disorders; severe injection-related infections; randomized controlled trial; hospital-based care; harm reduction
MeSH Terms: conditions — Substance-Related Disorders; Harm Reduction | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: The study will recruit patients at bedside in the hospital setting at approximately six hospitals and randomly assign approximately 480 inpatients in 1:1 ratio to the SIRI Team vs. TAU. Randomization will be stratified by 1) hospital site, 2) primary drug (opioid versus non-opioid), and 3) admission to intensive care unit (ICU) as part of the index hospitalization (ICU versus non-ICU) as a proxy for severity of infection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SIRI Team (Experimental): The study intervention ("SIRI Team") consists of a hospital-based multidisciplinary (ID/SUD consult) team that will provide intensive, integrated care for participants' ID and SUD both during the hospital stay and post-discharge for up to four months post-randomization. The SIRI Team will provide low barrier access to medications and harm reduction services for SUD; streamline ID/SUD treatment; provide longitudinal care with familiar providers; leverage different areas of expertise between physicians, advance practice providers, and patient navigators; and create patient-centered treatment plans, tailored to the individual, and informed by each patient's social circumstances, substance use, and personal goals/desires.
  Interventions: Behavioral: SIRI Team
- Treatment as Usual (Active Comparator): Treatment as Usual (TAU) will consist of the current healthcare landscape at each participating hospital site.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: SIRI Team — Participants randomized to the intervention will receive integrated ID and SUD care (SIRI Team) both during the hospitalization and after hospital discharge for 4 months post-randomization. The intervention is based upon six general principles for treating PWID with infectious complications and is informed by harm reduction.
  1. Medications for SUD as integral to management of infectious complications
  2. Integration of ID and SUD care
  3. Longitudinal care with familiar providers
  4. Multidisciplinary care and care coordination
  5. Tailored antibiotic options and care settings
  6. Harm reduction
  Arms: SIRI Team
Behavioral: Treatment as Usual — Participants assigned to the TAU group will receive the standard treatment for their severe injection-related infection and substance use disorder at each hospital. While TAU may differ between sites, it is typically comprised of a patient being cared for primarily by a hospital medicine physician (hospitalist) with consultation by infectious diseases (ID) and either psychiatry or addiction medicine physician. If the ID or addiction teams believe post-hospitalization follow up is indicated, each service will follow local protocols for arranging post-discharge continuation of care.
  Arms: Treatment as Usual

SUMMARY:
The goal of this clinical trial is to test the effectiveness of an integrated infectious disease/substance use disorder (SUD) clinical team intervention approach in patients hospitalized with severe injection-related infections (SIRI) who use drugs. The main question this study aims to answer is whether this intervention approach will be associated with lower mortality and fewer hospital readmissions. Participants will participate in the integrated SUD/ID care team intervention (SIRI Team). Researchers will compare this intervention to treatment as usual (TUA) to see if there are any differences in health outcomes.

DETAILED DESCRIPTION:
The study intervention ("SIRI Team") consists of a hospital-based multidisciplinary (ID/SUD consult) team that will provide intensive, integrated care for participants' ID and SUD both during the hospital stay and post-discharge for up to four months post-randomization. The SIRI Team will provide low barrier access to medications and harm reduction services for SUD; streamline ID/SUD treatment; provide longitudinal care with familiar providers; leverage different areas of expertise between physicians, advance practice providers, and patient navigators; and create patient-centered treatment plans, tailored to the individual, and informed by each patient's social circumstances, substance use, and personal goals/desires. The SIRI Team intervention will be grounded in a harm reduction approach. The intervention duration is approximately 4 months. Participants will complete follow-up visits at 4-, 8-, and 12-months post-randomization.

ELIGIBILITY:
Inclusion Criteria:

* Be admitted to a participating hospital at the time of randomization
* Be 18 years of age or older
* Currently be experiencing a severe injection-related infection/SIRI or suspected SIRI
* Have an indication of injecting drugs in the prior year
* Provide informed consent
* Ability to communicate in English
* Provide sufficient locator information
* Sign a HIPAA form and/or EHR release to facilitate record abstraction
* Report being willing to return for follow-up visits

Exclusion Criteria:

All individuals meeting any of the exclusion criteria will be excluded from study participation. Specifically, individuals will be excluded from participation if they:

* have significant cognitive or developmental impairment to the extent that they are unable to provide informed consent
* (or their legal guardian/representative) are unable or unwilling to give written informed consent
* are currently in jail, prison or other overnight facility as required by court of law or have pending legal action that could prevent participation in study activities
* are terminated via site principal investigator decision with agreement from one of the study lead investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2027-04-03 (Estimated); Study Completion 2027-04-03 (Estimated)

PRIMARY OUTCOMES:
Mortality and Hospital Readmissions | 4 months post-randomization
  Binary: A participant is alive with no hospital readmission 4 months post-randomization vs. a participant has died or been readmitted to the hospital within 4 months post-randomization

SECONDARY OUTCOMES:
Initiation of treatment before hospital discharge | Course of hospital visit (expected to be within 1 month of randomization)
  Binary: If patient initiated any of the treatments listed in protocol vs. if they did not engage
Receipt of post-discharge treatment | This will be a repeated assessment at each of the follow-up times. The main test of the secondary hypothesis is at the 4th month. An additional contrast will assess if this maintains on average at the 8th and 12th month.
  Binary: If patient initiated any of the treatments listed in protocol vs. if they did not engage
Completion of planned antibiotic course for the index infection | Course of antibiotic treatment (Length varies by severity of infection); Assessed at the 4 month follow-up time
  Binary: If patient completed planned antibiotic course for the index infection vs. if they did not complete antibiotic course
Patient-directed discharge from index hospitalization | Course of hospital visit (expected to be within 1 month of randomization)
  Binary: Patient discharges themselves from the hospital prior to the attending physician's orders to discharge vs. does not discharge themselves
Post-discharge hospital visits | This will be a repeated assessment at each of the follow-up times. The main test of the secondary hypothesis is at the 4th month. An additional contrast will assess if this maintains on average at the 8th and 12th month.
  Count: # of post-discharge hospital visits using repeated measures across all 3 follow-up visits
New or recurrent acute bacterial or fungal infection post-index hospitalization | This will be a repeated assessment at each of the follow-up times. The main test of the secondary hypothesis is at the 4th month. An additional contrast will assess if this maintains on average at the 8th and 12th month.
  Binary: Participant has a recurrent or persistent acute bacterial or fungal infection during the period of assessment vs. does not have a recurrent or persistent acute bacterial or fungal infection
Substance use severity | The main test of the secondary hypothesis is at the 4th month. An additional contrast will assess if this maintains on average at the 8th and 12th month.
  Continuous: Assessed via Drug Abuse Screening Test (DAST-10) scale; Range of scores [0 - 10], higher scores indicate worse outcome
Alcohol use severity | The main test of the secondary hypothesis is at the 4th month. An additional contrast will assess if this maintains on average at the 8th and 12th month.
  Continuous: Assessed via Alcohol Use Disorders Identification Test (AUDIT) scale; Range of scores [0 - 40], higher scores indicate worse outcome
All-cause mortality | At each of the follow-up times (4, 8 and 12 months)
  Binary: Mortality from all causes at any of the follow-up timepoints vs. alive at all timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Lisa R Metsch, PhD, Principal Investigator — Columbia University; David P Serota, MD, MSc, Principal Investigator — University of Miami; Daniel J Feaster, PhD, Principal Investigator — University of Miami; Carlos del Rio, MD, Principal Investigator — Emory University
Locations (6):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Miami - Jackson Memorial Hospital, Miami, Florida
  - Tampa General Hospital, Tampa, Florida
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Utah Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Information about the study and the de-identified study data will be available at https://datashare.nida.nih.gov/ within 18 months of the date the data are locked, as per the procedures of the National Drug Abuse Treatment Clinical Trials Network.
Time Frame: Within 18 months
Access Criteria: Information will be de-identified.
URL: https://datashare.nida.nih.gov/